CLINICAL TRIAL: NCT00084253
Title: Phase IV Study of Boosted Atazanavir (ATV) Versus Non-boosted ATV in Naive Patients
Brief Title: Study of Boosted Atazanavir (ATV) Versus Non-boosted ATV in Naive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-089 ST
Record Dates: First submitted 2004-06-09; First posted 2004-06-11 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Lamivudine; atazanavir, ritonavir drug combination

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Atazanavir/ Stavidine / Lamivudine
- 2 (Active Comparator)
  Interventions: Drug: Atazanavir-Ritonavir/ Stavidine / Lamivudine

INTERVENTIONS:
Drug: Atazanavir/ Stavidine / Lamivudine — Capsules, Oral, ATV (2 x 200 mg) QD + 3TC (2 x 150 mg) QD + Zerit XR (1 x 100 mg) QD, Once daily, 96 weeks.
  Other Names: Reyataz
  Arms: 1
Drug: Atazanavir-Ritonavir/ Stavidine / Lamivudine — Capsules, Oral, ATV (2 x 150 mg) QD + RTV (1 x 100 mg) QD + 3TC (2 x 150 mg) QD + Zerit XR (1 x 100 mg) QD*, Once daily, 96 weeks.
  Other Names: Reyataz
  Arms: 2

SUMMARY:
The purpose of this study is to find out if 300 mg of ATV plus 100 mg of ritonavir (RTV) works as well as 400 mg of ATV alone as part of a regimen with stavudine XR and lamivudine to slow or stop the progression of HIV infection in patients who have never used anti-HIV drugs.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* HIV RNA greater than or equal 200 copies/mL at screening
* 18 years old or older
* Must use barrier contraception
* Women of child-bearing potential must have a negative serum or urine pregnancy test within 72 hours before beginning to take the study medications

Exclusion Criteria:

* Unable or unwilling to use acceptable method of birth control for the entire study period including 8 weeks after the study
* Women using oral contraceptives, pregnant or breastfeeding women
* Women who have a positive pregnancy test on enrollment or before beginning to take the study medications
* People who have a life expectancy of greater than 12 months
* Newly diagnosed HIV-related OI or any medical condition requiring acute therapy at the time of enrollment
* Any antiretroviral therapy within 30 days prior to screening
* Any prior antiretroviral therapy (greater than 30 days of NRTI and/or greater than 7 days of non-nucleoside reverse-transcriptase inhibitor (NNRTI) or protease inhibitor therapies)
* Any of the following conditions: Cushings Syndrome, Gilbert's Syndrome, untreated hypothyroidism or hyperthyroidism, suspected primary (acute) HIV infection, obstructive liver disease, proven or suspected acute hepatitis in the 30 days prior to study entry, Intractable diarrhea (at greater than 6 loose stools per day for at least 78 consecutive days) within 30 days prior to study entry, history of hemophilia, history of acute or chronic pancreatitis, presence of cardiomyopathy (due to any cause) or any significant cardiovascular disease, such as unstable ischemic heart disease
* Active alcohol or substance abuse
* History or signs and symptoms of bilateral peripheral neuropathy greater than grade 2 at the time of screening
* Previous therapy with myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 3 months of study start or the expected need for such therapy or therapy with methadone or ribavirin/interferons or treatment with neurotoxic drugs or drugs that affect CYP3A4
* Inability to swallow capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-06; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To compare the proportion of subjects responding to treatment with HIV RNA levels < LOQ (400 c/mL) through Week 48 in treatment naive subjects for ATV and ATV/RTV (each combined with 3TC and d4T XR).

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Various locations within the US, Call For Information, New Jersey, United States